CLINICAL TRIAL: NCT05577156
Title: Sexual Quality of Life and Metastatic Breast Cancer
Brief Title: SexoMBC2 Non Interventional Study
Acronym: SexoMBC2
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01192-41
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Quality of Life; Sexual Behavior
MeSH Terms: conditions — Breast Neoplasms; Sexual Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Behavioral: Self-questionnaires and semi-structured interview

INTERVENTIONS:
Behavioral: Self-questionnaires and semi-structured interview — Patients will fill these questionnaires : BISF-W, QLQ-C30, QLQ-BR23 and if they agree answer to a semi-structured interview composed of 5 questions

SUMMARY:
The study is composed of three paper self-questionnaires to be filled in by the patients included at distance (> 6 months) from their diagnosis of metastatic breast cancer, in order to limit the impact of the announcement on the filling out the questionnaires.

After verification of the eligibility criteria, the medical oncologist will present the study to patients coming to the ICL for a follow-up consultation as part of their regular care. The patients will meet with a clinical research nurse so that she can explain the again and answer any questions they may have. She will also give the patients the questionnaires questionnaires and will give a presentation of the questions asked. After this meeting, the patients will be given sufficient time to reflect on, which may extend until their next visit to the ICL, in order to express, if they wish, their opposition to participating in the study. If she agrees to participate, the patient can then complete the questionnaires as well as the complementary questionnaire and place them in a closed envelope to be given to the clinical research nurse. The completion of the questionnaires will be completely anonymous. The data of those who object to the use of their data will be deleted from the database.

After the completion of the questionnaires, and in order to allow a benefit for the patient, a semi-directive interview in the form of a teleconsultation with a psycho-oncologist and sexologist will be offered. The interviews are not mandatory.

The time to fill in the self-questionnaires is estimated at 30 minutes and the semi-directive interview can last up to one hour. Finally, at the end of the study, as part of her subsequent care, each patient participating in the study will have the possibility to renew a teleconsultation with the psycho-oncologist and sexologist if she feels the need. As the subject of the study may generate personal questions and lead to a request for psychological and/or sexological care.

ELIGIBILITY:
Inclusion Criteria:

* Major woman
* Patient with metastatic breast cancer, either initially or secondary metastatic breast cancer
* RH+/HER2- tumor
* Patient starting first line metastatic therapy or currently undergoing 1st line metastatic treatment
* Patient diagnosed with metastatic breast cancer 6 months or more
* WHO 1 or 2 patient
* Postmenopausal or not
* Patient able to understand the French language

Exclusion Criteria:

* Patient WHO>2
* Patient undergoing chemotherapy
* HER2+ or triple negative tumor
* Male
* Patient diagnosed with breast cancer less than 6 months ago
* Patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: this study is proposed to adult women with metastatic HR+/HER2- breast cancer in first-line treatment
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Assessment of sexual quality of life in women with HR+/HER2- metastatic breast cancer in first-line treatment | Day 0
  Patients will fill the questionnaire : BISF-W (Brief Index of Sexual Function for Women)

SECONDARY OUTCOMES:
Assessment of overall quality of life in women with HR+/HER2- metastatic breast cancer in first-line treatment | Day 0
  Patients will fill the QLQ-C30 questionnaire
Assessment of overall quality of life in women with HR+/HER2- metastatic breast cancer in first-line treatment | Day 0
  Patients will fill the QLQ+BR23 questionnaire
Assessment of sexual and emotional intimacy | Day 0
  semi-structured interview composed of 5 questions

CONTACTS AND LOCATIONS:
Overall Officials: VINCENT MASSARD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France